CLINICAL TRIAL: NCT01606137
Title: A Long-term, Open Label, Safety and Tolerability Study of Cannabis Based Medicine Extract in Patients Who Have Participated in a GW Clinical Study Using Cannabis Based Medicine.
Brief Title: A Study of the Long-term Safety of Sativex Use
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWEXT0102
Record Dates: First submitted 2012-05-21; First posted 2012-05-25 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis; Spasticity; Pain
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity; Pain | interventions — nabiximols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GW-1000-02 (Experimental): Active treatment
  Interventions: Drug: GW-1000-02

INTERVENTIONS:
Drug: GW-1000-02 — Contained delta-9-tetrahydrocannabinol (THC) (27 mg/ml) and cannabidiol (CBD) (25 mg/ml) as extract of Cannabis sativa L., with peppermint oil, 0.05% (v/v), in ethanol:propylene glycol (50:50) excipient. Each 100 μl actuation of the pump action spray delivered 2.7 mg THC and 2.5 mg CBD. A maximum daily exposure of 130 mg THC was specified by the UK regulatory authority authorisation.
  Other Names: Sativex

SUMMARY:
Subjects who had previously received GW-1000-02 in a GW study who opted to continue using it in the long-term were monitored for ongoing tolerability and evidence of clinical benefit.

DETAILED DESCRIPTION:
Subjects who had previously participated in a placebo controlled GW clinical study were screened and if eligible began dosing with GW-1000-02. Subjects were reviewed for tolerability and evidence of clinical benefit at weeks two and four and then every eight weeks. Subjects self-titrated to symptom resolution or maximum tolerated/allowable dose of 130 mg THC and 120 mg CBD.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent.
* Male or female aged 18 years or above.
* Diagnosed with a condition categorised as one of the following: multiple sclerosis, spinal cord conditions, peripheral nerve injury or central nervous system damage associated with vascular, traumatic, infective, genetic or metabolic disease and whose symptom(s) were not wholly relieved by currently available therapy, prior to the previous study of GW-1000-02 or placebo.
* Had participated in a GW clinical study using GW-1000-02 within the previous month.
* Had shown tolerability to the study medication during the previous GW study.
* Was expected, by the investigator, to gain clinical benefit from receiving long-term GW-1000-02.
* Were willing, if female and of child bearing potential or male subjects with a partner of child bearing potential, to ensure that effective contraception was used during the study and for three months thereafter.
* Had not used cannabinoids (cannabis, Marinol or Nabilone) for at least seven days before Visit 1 (the exception being GW-1000-02 given as study medication) and were willing to abstain from any use of cannabis during the study.
* Recent (within seven days) haematology and blood chemistry that was normal or considered clinically acceptable in view of the subjects underlying condition.
* Able (in the investigators opinion) and willing to comply with all study requirements.
* Willing for the Home Office to be notified of his or her participation in the study.
* Willing to allow his or her general practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* History of serious psychiatric illness, including schizophrenia, other psychotic illness or severe personality disorder other than depression associated with the underlying condition.
* Known or strongly suspected of alcohol or substance abuse or considered by the investigator to have been at risk of alcohol or substance abuse.
* Severe cardiovascular disorder, such as ischaemic heart disease, arrhythmias (other than well controlled atrial fibrillation), poorly controlled hypertension or severe heart failure.
* History of epilepsy or convulsions.
* Significant renal or hepatic impairment.
* Terminally ill.
* Any other significant disease or disorder which, in the opinion of the investigator, may have either put the subject at risk because of participation in the study, or may have influenced the result of the study, or the subject's ability to participate in the study.
* Female subjects who were pregnant, lactating or planning pregnancy during the course of the study.
* Regular levodopa (Sinemet, Sinemet Plus, Levodopa, L-dopa, Madopar, Benserazide) therapy within seven days of study entry.
* Known or suspected hypersensitivity to cannabinoids or any of the excipients of the study medication.
* Known or suspected adverse reaction to cannabinoids.
* Donation of blood during the study.
* Previous participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2002-02; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Serpell, ChB FRCA, Principal Investigator — Gartnavel General Hospital
Locations (1):
- Gartnavel General Hospital, Glasgow, United Kingdom

REFERENCES:
- [Result] Serpell MG, Notcutt W, Collin C. Sativex long-term use: an open-label trial in patients with spasticity due to multiple sclerosis. J Neurol. 2013 Jan;260(1):285-95. doi: 10.1007/s00415-012-6634-z. Epub 2012 Aug 10. PMID 22878432

RESULTS

PARTICIPANT FLOW:
Groups:
- GW-1000-02: Each actuation of oromucosal spray delivers 2.7mg delta-9-tetrahydrocannabinol (THC) and 2.5mg cannabidiol (CBD). The maximum permitted dose of was eight actuations in any three hour period, and 48 actuations in any 24 hour period (THC 130 mg : CBD 120 mg).
Period: Overall Study
Arm/Group | GW-1000-02
Started | 507
Completed | 245
Not Completed | 262
Not completed — Adverse Event | 85
Not completed — Withdrawal by Subject | 74
Not completed — Lack of Efficacy | 56
Not completed — Lost to Follow-up | 15
Not completed — Protocol Violation | 1
Not completed — Patient non-compliance | 9
Not completed — Death | 1
Not completed — Decreased/no pain | 4
Not completed — Issues with driving | 4
Not completed — multiple sclerosis less stable | 1
Not completed — Increased bilirubin | 1
Not completed — Spray causes nausea | 1
Not completed — Not enough improvement | 4
Not completed — Wanted to try another treatment | 1
Not completed — Patient leaving country | 1
Not completed — Personal reasons | 1
Not completed — Unable to tolerate study med. taste | 1
Not completed — Patient moving | 1
Not completed — Unable to collect consistent data | 1

BASELINE CHARACTERISTICS:
Arm/Group | GW-1000-02
Number analyzed (Participants) | 507
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 458
  >=65 years | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 288
  Male | 219
Region of Enrollment [Number; unit: participants]
  United Kingdom | 507

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events as a Measure of Subject Safety.
Description: Following data entry, all adverse events were medically encoded using the Medical Dictionary for Regulatory Activities (MedDRA) 6.0. All subjects who experienced an adverse event during the treatment period is presented.
Time Frame: Up to 1051 days
Population: All subjects who took part in the extension study were included in the analysis.
Measure: Number; unit: participants
Groups:
- GW-1000-02: Each 100 ul actuation contains 27 mg THC and 25 mg CBD. A maximum of 48 actuations (130 mg of THC 120 and mg of CBD) was permitted in any 24 hour period.
Arm/Group | GW-1000-02
Number analyzed (Participants) | 507
participants | 477

2. Secondary Outcome: Change From Parent Study Baseline in Spasticity 0-10 Numerical Rating Scale Score After 52 Weeks of Treatment.
Description: Subjects were asked to rate the severity of their primary symptom each week in the diary using an 11-point Numerical Rating Scale, where zero = "best possible" and 10 = "worst possible". A negative value indicates an improvement in score from baseline.
Time Frame: 0 - 52 weeks
Population: All subjects who entered the study from a parent randomised controlled trial (RCT) investigating the efficacy of GW-1000-02 in the treatment of spasticity associated with multiple sclerosis, and who received at least one actuation of study medication were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02
Number analyzed (Participants) | 61
units on a scale | -1.83 (2.41)

3. Secondary Outcome: Change From Parent Study Baseline in Central Neuropathic Pain 0-10 Numerical Rating Scale Score at 52 Weeks of Treatment.
Description: as for outcome 2
Time Frame: 0 - 52 weeks.
Population: All subjects who entered the study from a central neuropathic pain parent RCT and received at least one actuation of study medication were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02
Number analyzed (Participants) | 62
units on a scale | -2.96 (2.03)

4. Secondary Outcome: Change From Parent Study Baseline in Neuropathic Pain 0-10 Numerical Rating Scale Score at 52 Weeks of Treatment in Multiple Sclerosis Subjects.
Description: as for outcome 2
Time Frame: 0 - 52 weeks.
Population: All subjects who entered the study from a neuropathic pain in multiple sclerosis parent RCT and received at least one actuation of study medication were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02
Number analyzed (Participants) | 63
units on a scale | -3.11 (1.90)

5. Secondary Outcome: Change From Parent Study Baseline in Pain 0-10 Numerical Rating Scale Score at 52 Weeks of Treatment.
Description: as for outcome 2
Time Frame: 0 - 52 weeks.
Population: All subjects who entered the study from a pain parent RCT and received at least one actuation of study medication were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GW-1000-02
Number analyzed (Participants) | 131
units on a scale | -2.57 (2.02)

6. Secondary Outcome: Subject Assessment of Benefit at the Last Study Visit in Those Experiencing Neuropathic Pain Due to Multiple Sclerosis.
Description: Assessment of benefit achieved at study completion/withdrawal was evaluated by the subject, and the number of subjects who perceived a benefit from treatment is presented.
Time Frame: Up to 1051 days
Population: All multiple sclerosis subjects who entered the study from a neuropathic pain parent RCT and received at least one actuation of study medication were included in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | GW-1000-02
Number analyzed (Participants) | 98
participants | 75

7. Secondary Outcome: Investigator Assessment of Benefit at the Last Study Visit in Those Experiencing Neuropathic Pain Due to Multiple Sclerosis.
Description: Assessment of benefit achieved at study completion/withdrawal was evaluated by the investigator, and the number of subjects that investigators considered to have experienced a benefit from the treatment is presented.
Time Frame: Up to 1051 days
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | GW-1000-02
Number analyzed (Participants) | 98
participants | 76

8. Secondary Outcome: Subject Assessment of Benefit at the Last Study Visit in Those Experiencing Central Neuropathic Pain.
Description: as for outcome 6
Time Frame: Up to 1051 days
Population: All subjects who entered the study from a neuropathic pain parent RCT and received at least one actuation of study medication were included in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | GW-1000-02
Number analyzed (Participants) | 168
participants | 112

9. Secondary Outcome: Investigator Assessment of Benefit at the Last Study Visit in Those Experiencing Central Neuropathic Pain.
Description: as for outcome 7
Time Frame: Up to 1051days
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | GW-1000-02
Number analyzed (Participants) | 168
participants | 111

10. Secondary Outcome: Subject Assessment of Benefit at the Last Study Visit in Those Experiencing Pain.
Description: as for outcome 6
Time Frame: Up to 1051
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | GW-1000-02
Number analyzed (Participants) | 314
participants | 193

11. Secondary Outcome: Investigator Assessment of Benefit at the Last Study Visit in Those Experiencing Pain.
Description: as for outcome 7
Time Frame: Up to 1051 days
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | GW-1000-02
Number analyzed (Participants) | 314
participants | 190

12. Secondary Outcome: Subject Assessment of Benefit at the Last Study Visit in All Multiple Sclerosis Subjects.
Description: as for outcome 6
Time Frame: Up to 1051 days
Population: All subjects who entered the study from a multiple sclerosis parent RCT and received at least one actuation of study medication were included in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | GW-1000-02
Number analyzed (Participants) | 286
participants | 199

13. Secondary Outcome: Investigator Assessment of Benefit at the Last Study Visit in All Multiple Sclerosis Subjects.
Description: as for outcome 7
Time Frame: Up to 1051 days.
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | GW-1000-02
Number analyzed (Participants) | 287
participants | 200

14. Secondary Outcome: Investigator Global Assessment at the Last Study Visit in Subjects With Neuropathic Pain Due to Multiple Sclerosis.
Description: Investigators rated the global severity of the subject's underlying primary condition, e.g. their MS or spinal cord injury, since the previous visit using a five point scale of "much worse", "worse", "no change", "better", "much better". The number of subjects rated by the investigator as "better" or "much better" at the last study visit is presented.
Time Frame: Up to 1051 days
Population: All subjects who entered the study from a parent RCT investigation neuropathic pain due to multiple sclerosis, and who received at least one actuation of study medication were included in the efficacy analysis.
Measure: Number; unit: participants
Arm/Group | GW-1000-02
Number analyzed (Participants) | 98
participants | 30

15. Secondary Outcome: Investigator Global Assessment at the Last Study Visit in Subjects With Central Neuropathic Pain.
Description: as for outcome 14
Time Frame: Up to 1051 days.
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | GW-1000-02
Number analyzed (Participants) | 166
participants | 83

16. Secondary Outcome: Investigator Global Assessment at the Last Study Visit in Subjects With Pain.
Description: as for outcome 14
Time Frame: Up to 1051 days.
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | GW-1000-02
Number analyzed (Participants) | 312
participants | 122

17. Secondary Outcome: Investigator Global Assessment at the Last Study Visit in Subjects With Multiple Sclerosis.
Description: as for outcome 14
Time Frame: Up to 1051 days.
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | GW-1000-02
Number analyzed (Participants) | 284
participants | 87

ADVERSE EVENTS:
Time Frame: All adverse events occurring from the extension study onset to the last study visit (up to 1051 days) were collected. All deaths and serious adverse events occurring within 28 days of the final dose of study medication were also collected.
Description: All adverse events occurring during the study were reported on the running logs at the back of the study case report form.
Arm/Group | GW-1000-02
Serious Adverse Events (participants affected / at risk) | 74/507
Other Adverse Events (participants affected / at risk) | 477/507
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GW-1000-02 (N=507)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1
VENTRICULAR BIGEMINY (Cardiac disorders) | 1
CORNEAL ULCER (Eye disorders) | 1
EYELID OEDEMA (Eye disorders) | 1
ABDOMINAL PAIN NOT OTHERWISE SPECIFIED (NOS) (Gastrointestinal disorders) | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2
DIARRHOEA NOS (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2
VOMITING NOS (Gastrointestinal disorders) | 2
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1
CONSTIPATION AGGRAVATED (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 1
HAEMATEMESIS (Gastrointestinal disorders) | 1
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1
OESOPHAGITIS NOS (Gastrointestinal disorders) | 1
SMALL INTESTINAL GANGRENE NOS (Gastrointestinal disorders) | 1
SMALL INTESTINAL OBSTRUCTION NOS (Gastrointestinal disorders) | 1
CHEST PAIN (General disorders) | 2
WEAKNESS (General disorders) | 2
PAIN EXACERBATED (General disorders) | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 1
DRUG HYPERSENSITIVITY (Immune system disorders) | 2
URINARY TRACT INFECTION NOS (Infections and infestations) | 14
SEPSIS NOS (Infections and infestations) | 2
BRONCHOPNEUMONIA NOS (Infections and infestations) | 1
CELLULITIS (Infections and infestations) | 1
GASTROENTERITIS NOS (Infections and infestations) | 1
INFECTION NOS (Infections and infestations) | 1
KLEBSIELLA SEPSIS (Infections and infestations) | 1
LOWER RESPIRATORY TRACT INFECTION NOS (Infections and infestations) | 1
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 1
PNEUMONIA NOS (Infections and infestations) | 1
POST PROCEDURAL SITE WOUND INFECTION (Infections and infestations) | 1
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 2
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1
DEVICE FAILURE (Injury, poisoning and procedural complications) | 1
FRACTURED PELVIS NOS (Injury, poisoning and procedural complications) | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1
INCISIONAL HERNIA NOS (Injury, poisoning and procedural complications) | 1
MEDICAL DEVICE COMPLICATION (Injury, poisoning and procedural complications) | 1
POST PROCEDURAL URINE LEAK (Injury, poisoning and procedural complications) | 1
LIVER FUNCTION TESTS NOS ABNORMAL (Investigations) | 2
BLOOD IN STOOL (Investigations) | 1
WEIGHT DECREASED (Investigations) | 1
HYPOGLYCAEMIA NOS (Metabolism and nutrition disorders) | 2
ANOREXIA (Metabolism and nutrition disorders) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
INGUINAL MASS (Musculoskeletal and connective tissue disorders) | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1
LUNG CANCER STAGE UNSPECIFIED (EXCL METASTATIC TUMOURS TO LUNG) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 5
MULTIPLE SCLEROSIS AGGRAVATED (Nervous system disorders) | 4
CONVULSIONS NOS (Nervous system disorders) | 2
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 2
DIZZINESS (Nervous system disorders) | 2
DYSARTHRIA (Nervous system disorders) | 2
SOMNOLENCE (Nervous system disorders) | 2
GRAND MAL CONVULSION (Nervous system disorders) | 1
HYPOAESTHESIA (Nervous system disorders) | 1
PARAESTHESIA (Nervous system disorders) | 1
TREMOR (Nervous system disorders) | 1
SUICIDAL IDEATION (Psychiatric disorders) | 2
DELUSIONAL PERCEPTION (Psychiatric disorders) | 1
PARANOIA (Psychiatric disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 2
RENAL FAILURE ACUTE ON CHRONIC (Renal and urinary disorders) | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1
URTICARIA NOS (Skin and subcutaneous tissue disorders) | 1
PREGNANCY OF PARTNER (Social circumstances) | 4
CIRCULATORY COLLAPSE (Vascular disorders) | 1
DEEP VENOUS THROMBOSIS NOS (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GW-1000-02 (N=507)
Dizziness (Nervous system disorders) | 144
Headache Not Otherwise Specified (NOS) (Nervous system disorders) | 56
Somnolence (Nervous system disorders) | 43
Dysgeusia (Nervous system disorders) | 39
Multiple Sclerosis Aggravated (Nervous system disorders) | 39
Multiple Sclerosis Relapse (Nervous system disorders) | 30
Balance Impaired NOS (Nervous system disorders) | 27
Memory Impairment (Nervous system disorders) | 18
Disturbance in Attention (Nervous system disorders) | 17
Nausea (Gastrointestinal disorders) | 87
Diarrhoea NOS (Gastrointestinal disorders) | 60
Vomiting NOS (Gastrointestinal disorders) | 55
Dry Mouth (Gastrointestinal disorders) | 43
Mouth Ulceration (Nervous system disorders) | 28
Constipation (Gastrointestinal disorders) | 27
Glossodynia (Gastrointestinal disorders) | 26
Oral Pain (Gastrointestinal disorders) | 24
Dyspepsia (Gastrointestinal disorders) | 23
Tooth Discolouration (Gastrointestinal disorders) | 19
Fatigue (General disorders) | 61
Weakness (General disorders) | 34
Fall (General disorders) | 26
Pain Exacerbated (General disorders) | 25
Feeling Drunk (General disorders) | 25
Application Site Pain (General disorders) | 24
Lethargy (General disorders) | 18
Oedema Peripheral (General disorders) | 17
Influenza Like Illness (General disorders) | 16
Malaise (General disorders) | 16
Urinary Tract Infection NOS (Infections and infestations) | 111
Nasopharyngitis (Infections and infestations) | 40
Lower Respiratory Tract Infection NOS (Infections and infestations) | 30
Influenza (Infections and infestations) | 19
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 35
Arthralgia (Musculoskeletal and connective tissue disorders) | 31
Back Pain (Musculoskeletal and connective tissue disorders) | 27
Pain in Limb (Musculoskeletal and connective tissue disorders) | 24
Euphoric Mood (Psychiatric disorders) | 22
Depression (Psychiatric disorders) | 20
Depressed Mood (Psychiatric disorders) | 18
Insomnia (Psychiatric disorders) | 18
Anxiety (Psychiatric disorders) | 15
Gamma-glutamyltransferase Increased (Investigations) | 26
Weight Decreased (Investigations) | 20
Alanine Aminotransferase Increased (Investigations) | 16
Blood Alkaline Phosphatase NOS Increased (Investigations) | 13
Contusion (Skin and subcutaneous tissue disorders) | 16
Rash NOS (Skin and subcutaneous tissue disorders) | 16
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GW will coordinate the dissemination of data from this study and may solicit input and assistance from the principal investigator. All publications, for example manuscripts, abstracts, oral/slide presentations or book chapters based on this study, must be submitted to GW for corporate review before release.